CLINICAL TRIAL: NCT02695290
Title: An Open-label, Single-arm Phase IV Study of Afatinib in Patients With Stage IV or Recurrent Non-Small Cell Lung Cancer Who Have Poor Performance Status and Whose Tumors Have the Common Epidermal Growth Factor Receptor (EGFR) Mutations, Exon 19 Deletions or Exon 21(L858R) Substitution Mutations
Brief Title: Afatinib in EGFR+NSCLC (Recurrent or Stage IV) - Patients With Poor Performance Status (ECOG 2 or 3)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.208
Record Dates: First submitted 2016-02-25; First posted 2016-03-01 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung; ErbB Receptors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

ARMS (1):
- Afatinib (Experimental)
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib

SUMMARY:
There is a medical need for improving treatment of poor performance status patients with EGFR driver mutations and documenting safety and tolerability of existing agents.

ELIGIBILITY:
Inclusion criteria:

* Pathologically or cytologically confirmed NSCLC
* Stage IV Cancer (includes cytologically proven pleural effusion or pericardial effusion) or recurrent disease. The staging is based on American Joint Committee on Cancer (AJCC) Tumor Node Metastatic (TNM) classification of malignant tumors, 7th edition
* Evidence of common EGFR activating mutations (Del 19 and/or L858R)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 2 or 3
* Adequate organ function, defined as all of the following:
* Absolute neutrophil count (ANC) > 1500 / mm3
* Platelet count >75,000 / mm3.
* Baseline creatinine of < or = 1.5 g/dl or, if > 1.5, an estimated creatinine clearance of > 45 ml/min
* Total Bilirubin < 1.5 times upper limit of institutional normal (ULN)
* Aspartate amino transferase (AST) or alanine amino transferase (ALT) < three times ULN (if related to liver metastases < five times ULN)
* Recovery from any previous therapy related toxicity to< or = Grade 1 at study entry (except for stable sensory neuropathy < or =Grade 2 and alopecia)
* Life expectancy of at least three months
* Written informed consent that is consistent with International Council on Harmonization- Good Clinical Practice (ICH-GCP) guidelines
* Age 18 or older

Exclusion criteria:

* Prior participation in an afatinib clinical study, even if not assigned to afatinib treatment
* Prior systemic therapy for metastatic or recurrent NSCLC including prior treatment with EGFR targeting small molecules or antibodies. Note: radiotherapy alone and adjuvant/neoadjuvant treatment is not counted as a line of therapy.
* Concurrent investigational therapy or investigational therapy within 4 weeks of start of afatinib therapy
* Radiotherapy within 4 weeks prior to start of study treatment, except as follows:

  i.) Palliative radiation to target organs other than chest may be allowed up to 2 weeks prior to study treatment, or ii.) Single dose palliative treatment (e.g Stereotactic Radio Surgery(SRS) or Stereotactic Body Radiation Therapy) (SBRT) for symptomatic metastasis outside above allowance to be discussed with sponsor prior to enrolling.
* Major surgery within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study
* Women of child-bearing potential (WOCBP) and men who are able to father a child, or use adequate contraception prior to study entry, for the duration of study participation and for at least 28 days after treatment has ended.
* Presence of an active infection or with a fever > 38.5 C within 3 days of the first scheduled day of dosing
* Known hypersensitivity to afatinib or the excipients of afatinib
* Known pre-existing interstitial lung disease
* Pathologically documented meningeal carcinomatosis (i.e. cytology (+) lumbar puncture ; radiology reports alone raising this as a possibility, in the absence of true symptomatology, would not constitute an exclusion)
* Presence of brain or subdural metastases, unless local therapy has been completed and use of corticosteroids has been discontinued or the dose has been stable for at least 4 weeks before starting study treatment. Any symptoms attributed to brain metastases must be stable for at least 4 weeks before starting study treatment (Pts post SRS can be enrolled earlier as long as their symptoms are stable or improved and they are off steroids)
* Previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 2 years and is considered to be cured
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New York Heart Association (NYHA) classification of 3 or 4 unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to treatment with afatinib.
* Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug (e.g. Crohn's disease, ulcerative colitis, chronic diarrhoea, malabsorption)
* Known or suspected active hepatitis B (Hep B) infection (defined as presence of HepB (surface Antigen) sAg and/ or Hep B DNA), active hepatitis C infection (defined as presence of Hep C RNA) and/or known HIV carrier
* Any history of or concomitant condition that, in the opinion of the Investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the safety and efficacy of the test drug
* Treatment with any of the prohibited concomitant medications that cannot be stopped for the duration of trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2016-08-26 (Actual); Study Completion 2016-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1200.208.10032 Boehringer Ingelheim Investigational Site, Fountain Valley, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, single-arm Phase IV study of afatinib in patients with stage IV or recurrent Non-Small Cell Lung Cancer who have poor performance status and whose tumors have the common epidermal growth factor receptor (EGFR) mutations, Exon 19 deletions or Exon 21(L858R) substitution mutations.
Groups:
- Afatinib: Subject received Giotrif® / Gilotrif® (Afatinib) with starting dose of 30 milligram (mg) orally, once daily until progression or occurrence of intolerable adverse event (AE) or end of trial.
Period: Overall Study
Arm/Group | Afatinib
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients who receive at least one dose of afatinib will be included in the treated set. All data collected from the single patient who received study medication.
Arm/Group | Afatinib
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62 (NA) — Not Applicable as only one patient was treated
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Occurrence of Adverse Events (AEs) Leading to Dose Reduction of Afatinib
Description: Percentage of patients with occurrence of Adverse Events (AEs) leading to dose reduction of afatinib.
Time Frame: Up to 98 days
Population: Patients who receive at least one dose of afatinib will be included in the treated set.All data collected from the single patient who received study medication.
Measure: Number (95% Confidence Interval); unit: Pecentage of Participants
Arm/Group | Afatinib
Number analyzed (Participants) | 1
Pecentage of Participants | 0.0 [NA to NA] — Confidence interval is not calculable as only one patient is analyzed.

2. Secondary Outcome: Percentage of Patients With Occurrence of CTCAE Grade 3 or Higher Diarrhoea, Rash/Acne+, Stomatitis+ and Paronychia+ (+ Represents Grouped Term)
Description: Percentage of patients with occurrence of Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher diarrhoea, rash/acne+, stomatitis+ and paronychia+ (+ represents grouped term).
Time Frame: Up to 98 days
Population: Patients who receive at least one dose of afatinib will be included in the treated set.All data collected from the single patient who received study medication. All data collected from the single patient who received study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Afatinib
Number analyzed (Participants) | 1
Percentage of Participants | 0

3. Secondary Outcome: Time to First Dose Reduction of Afatinib Caused by Adverse Events (AEs)
Description: Time to first dose reduction of afatinib caused by Adverse Events (AEs) defined as time from the date of the first administration of afatinib to the first dose reduction of afatinib caused by AEs.
Time Frame: Up to 98 days
Population: All data collected from the single patient who received study medication. As none of the AEs led to the dose reduction hence time to first dose reduction is not applicable.
Arm/Group | Afatinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first drug administration until 40 days after the last dose of study medication, up to 98 days
Arm/Group | Afatinib
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (N=1)
Diarrhoea (Gastrointestinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1

LIMITATIONS AND CAVEATS:
This study was stopped prematurely when only 1 patient had received afatinib treatment so it was not possible to draw any conclusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.